CLINICAL TRIAL: NCT01005342
Title: The Influence of Dietary Fibre-rich Meals on Gene Expression in Leukocytes and Postprandial Glucose and Lipid Response in Healthy Subjects
Brief Title: Influence of Dietary Fiber-rich Meals on Gene Expression and Postprandial Glucose and Lipid Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government); Oatly AB (Unknown); Lantmannen Food R&D (Unknown); Danisco Sugar AB/Fibrex (Unknown)
Responsible Party: Gunilla Önning, Lund University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: KCROS07
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Hypoglycemia; Hyperglycemia
Keywords: gene expression; oats; rye; sugar beet fiber; glucose; insulin; triglyceride; decreased postprandial glucose; decreased postprandial insulin; glycemic index
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia; Insulin Resistance | interventions — beta-Glucans; arabinoxylan; Sucrose; Pectins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Mixture of fiber (Experimental): Single intake of a mixture of spray-dried oat drink, rye bran and sugar beet fiber
  Interventions: Other: Mixture of fiber
- Sugar beet fiber (Experimental): Single intake of sugar beet fiber
  Interventions: Other: Sugar beet fiber
- Rye bran (Experimental): Single intake of rye bran
  Interventions: Other: Rye bran
- Oat bran (Experimental): Single intake of oat bran
  Interventions: Other: Oat bran
- Spray-dried oat drink (Experimental): Single intake of spray-dried oat drink
  Interventions: Other: Spray-dried oat drink
- Control (Placebo Comparator): Single intake of a meal with no added fiber
  Interventions: Other: Control

INTERVENTIONS:
Other: Oat bran — 82 g oat bran was added to 250 ml blackcurrant beverage with pulp to give 5 g soluble fiber (12.6 g total fiber).
  Other Names: Oats; Beta-glucan
  Arms: Oat bran
Other: Spray-dried oat drink — 62 g spray-dried oat drink was added to 250 ml blackcurrant beverage with pulp to give 2.7 g soluble fiber (3.3 g total fiber).
  Other Names: Oats; Oat milk; Beta-glucan
  Arms: Spray-dried oat drink
Other: Rye bran — 31 g rye bran was added to 250 ml blackcurrant beverage with pulp to give 1.7 g soluble fiber (12 g total fiber).
  Other Names: Rye; Arabinoxylan
  Arms: Rye bran
Other: Sugar beet fiber — 19 g sugar beet fiber was added to 250 ml blackcurrant beverage with pulp to give 5 g soluble fiber (12 g total fiber).
  Other Names: Sugar beet; Pectin
  Arms: Sugar beet fiber
Other: Mixture of fiber — 38 g spray-dried oat drink, 30 g rye bran and 6 g sugar beet fiber were added to 250 ml blackcurrant beverage with pulp to give 5 g soluble fiber (18 g total fiber).
  Arms: Mixture of fiber
Other: Control — No fiber was added to control meal (250 g black-currant beverage)
  Arms: Control

SUMMARY:
The aim of this study is to

* Measure the effect on gene expression in leukocytes from a meal rich in oat bran
* Investigate the postprandial glucose, insulin and triglyceride responses after intake of meals containing fiber from different sources (oat, rye and sugar beet fiber) or a meal containing a mixture of these three fibers

DETAILED DESCRIPTION:
Dietary fiber has long been known to give beneficial health effects. Yet, the understanding of how fiber-rich meals regulate molecular events at a gene level is limited. Also, few studies have compared the effects of different fiber sources on postprandial responses and hardly any study the effects of fiber mixtures in the same meal, even though this is more similar to regular eating habits.

Healthy subjects will come to the study center after an overnight fast, to ingest breakfasts randomly enriched with different fiber. The meals contains either spray-dried oat drink, rye bran, sugar beet fiber a mixture of these three fibers, oat bran or no added fiber (control). All meals are adjusted to contain the same total amount of available carbohydrates and fat. Blood leukocytes for gene expression profiling were taken before and 2 h after consumption while blood samples for analysis of postprandial glucose, insulin and triglyceride levels were taken every 30 min during 3 h.

NuGO Affymetrix Human Genechip NuGO_Hs1a520180 are used for the microarray analysis and analysis is performed with linear mixed models and enrichment analysis to identify functional gene sets that responded to the specific oat bran effect.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30

Exclusion Criteria:

* pregnancy
* breastfeeding
* diabetes mellitus
* hepatitis B
* blood lipid lowering pharmaceuticals
* intolerance or allergy to cereals or sugar beet fiber

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Changed gene expression profile by fiber-rich meals | 2 h after meal intake

SECONDARY OUTCOMES:
Lowering of postprandial glucose by fiber-rich meals | 0-180 min after meal intake

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Önning, Dr., Study Director — Lund University
Locations (1):
- Lund University, Lund, Sweden

REFERENCES:
- [Result] Ulmius M, Johansson A, Onning G. The influence of dietary fibre source and gender on the postprandial glucose and lipid response in healthy subjects. Eur J Nutr. 2009 Oct;48(7):395-402. doi: 10.1007/s00394-009-0026-x. Epub 2009 May 5. PMID 19415409